CLINICAL TRIAL: NCT00000691
Title: A Phase II Dose-Ranging, Open-Labelled Trial of Foscarnet Salvage Therapy for AIDS Patients With Sight-Threatening CMV Retinitis Who Cannot Be Treated With Ganciclovir Due To Myelosuppression or Treatment Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 093; 11068 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: Retinitis; AIDS-Related Opportunistic Infections; Ganciclovir; Drug Evaluation; Foscarnet; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome; Antiviral Agents
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; Retinitis; AIDS-Related Opportunistic Infections; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome | interventions — Foscarnet

INTERVENTIONS:
Drug: Foscarnet sodium

SUMMARY:
To examine the usefulness and safety of the antiviral drug foscarnet in treating AIDS patients with cytomegalovirus (CMV) infection that is causing sight-threatening inflammation of the retina in one or both eyes (CMV retinitis). Because of the seriousness of sight-threatening CMV retinitis in AIDS patients and a lack of other available treatments for those patients who cannot be treated with ganciclovir (DHPG) (because of its toxic effect on the body's blood-forming cells, because it did not control the disease, or because patient's blood cell or platelet counts are too low to begin with), it is worthwhile to try an immediate trial with foscarnet. AMENDED: ACTG 093 was originally designed as a randomized dose-ranging study of foscarnet maintenance therapy. Patients enrolled between March 17, 1989, and January 1, 1990, received either 60 mg/kg/day or 90/mg/kg day as maintenance therapy following the 2 week induction period. Based on the preliminary results of ACTG 015/915, which studied maintenance doses of foscarnet of 60 mg/kg/day, 90 mg/kg/day and 120 mg/kg/day, the 60-mg/kg/day and 90/mg/kg/day arms of this study have been closed. All patients entering the study beginning January 2, 1990 will receive foscarnet maintenance therapy on a 120/mg/kg/day algorithm following induction.

DETAILED DESCRIPTION:
Because of the seriousness of sight-threatening CMV retinitis in AIDS patients and a lack of other available treatments for those patients who cannot be treated with ganciclovir (DHPG) (because of its toxic effect on the body's blood-forming cells, because it did not control the disease, or because patient's blood cell or platelet counts are too low to begin with), it is worthwhile to try an immediate trial with foscarnet. AMENDED: ACTG 093 was originally designed as a randomized dose-ranging study of foscarnet maintenance therapy. Patients enrolled between March 17, 1989, and January 1, 1990, received either 60 mg/kg/day or 90/mg/kg day as maintenance therapy following the 2 week induction period. Based on the preliminary results of ACTG 015/915, which studied maintenance doses of foscarnet of 60 mg/kg/day, 90 mg/kg/day and 120 mg/kg/day, the 60-mg/kg/day and 90/mg/kg/day arms of this study have been closed. All patients entering the study beginning January 2, 1990 will receive foscarnet maintenance therapy on a 120/mg/kg/day algorithm following induction.

AMENDED: The ACTG 093 optional extended maintenance therapy period will conclude on January 2, 1991 in order to facilitate timely analysis of this study. All patients who wish to continue foscarnet therapy should be referred to Astra Protocol 90-FOS-14 at telephone number 800-292-5775. Original design: Patients are placed into two groups: (1) patients who have a sight-threatening lesion in the retina of an eye with vision that can be saved (corrected vision of 20/100 or better) and who cannot be treated with DHPG, and (2) patients whose retinitis has quickly gotten worse and/or has shown resistance to DHPG treatment. Both groups will receive a beginning (induction) dose of foscarnet by vein (IV) for 2 weeks, followed by a maintenance dose for 8 weeks with an option to continue up to 24 weeks. AMENDED: Patients entering the study on or after 01/02/90 receive the standard two week course of foscarnet induction therapy and receive maintenance therapy. Treatment is given for a ten week study period or until progression occurs or toxicity endpoints are reached. If retinitis is stable and foscarnet well-tolerated, maintenance therapy may be extended for a period not to exceed 1 year.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Aerosolized pentamidine for Pneumocystis carinii pneumonia (PCP) prophylaxis.
* Oral antibiotics if patient is hematologically stable on that regimen for at least 30 days prior to study entry.
* Therapy with vancomycin.
* Drug therapy for Kaposi's sarcoma if patient is hematologically stable for at least 30 days prior to study entry.
* Initiate or resume zidovudine (AZT) in 2nd week of foscarnet maintenance therapy at dose of 100 or 200 mg q4h at investigator's discretion.
* Initiate or continue erythropoietin therapy via the treatment IND mechanism.
* Initiate or continue therapy with investigational triazoles for disseminated fungal infections. Caution should be used in concurrent use of foscarnet and ciprofloxacin, as such use has appeared to exacerbate renal failure in one patient.

Prior Medication:

Allowed:

* Oral antibiotics if patient is hematologically stable on that regimen for at least 30 days prior to study entry.
* Drug therapy for Kaposi's sarcoma if patient is hematologically stable for at least 30 days prior to study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Corneal, lens, or vitreous opacification that precludes examination of the fundi.
* Clinically significant pulmonary or neurologic impairment, including intubation or coma.
* Karnofsky performance status = or < 50.

Concurrent Medication:

Excluded:

* Immunomodulators.
* Biologic response modifiers.
* Investigational agents (other than erythropoietin and investigational triazoles).
* Ganciclovir.
* Didanosine (ddI).
* Systemic acyclovir.
* CMV hyperimmune serum / globulin.
* Interferons.
* Nephrotoxic agents including aminoglycosides, amphotericin B, parenteral pentamidine.
* Caution should be used in the concurrent use of foscarnet and ciprofloxacin, as such use has appeared to exacerbate renal failure in one patient.

Patients with the following are excluded:

* Corneal, lens, or vitreous opacification that precludes examination of the fundi.
* Clinically significant pulmonary or neurologic impairment, including intubation or coma.
* Unwilling or unable to suspend zidovudine treatment until 2nd week of foscarnet maintenance therapy.

Prior Medication:

Excluded:

* Foscarnet for cytomegalovirus retinitis.
* Systemic acyclovir.
* Immunomodulators.
* Biologic response modifiers.
* Investigational agents (other than erythropoietin and investigational triazoles).

AIDS patients with active cytomegalovirus (CMV) retinitis who cannot be treated with ganciclovir. At least one pending CMV culture from both blood (buffy-coat) and urine must be obtained prior to study entry. Patients must be able to give informed consent. Patients with a history of a seizure disorder or central nervous system mass lesion will be included.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 156
Dates: Study Completion 1992-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MA Jacobson, Study Chair; C Crumpacker, Study Chair
Locations (11):
- United States (11):
  - USC CRS, Los Angeles, California
  - Ucsf Aids Crs, San Francisco, California
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Washington U CRS, St Louis, Missouri
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Cornell University A2201, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Duke Univ. Med. Ctr. Adult CRS, Durham, North Carolina

REFERENCES:
- [Background] Harb GE, Bacchetti P, Jacobson MA. Survival of patients with AIDS and cytomegalovirus disease treated with ganciclovir or foscarnet. AIDS. 1991 Aug;5(8):959-65. doi: 10.1097/00002030-199108000-00006. PMID 1663770
- [Background] Jacobson MA, Drew WL, Feinberg J, O'Donnell JJ, Whitmore PV, Miner RD, Parenti D. Foscarnet therapy for ganciclovir-resistant cytomegalovirus retinitis in patients with AIDS. J Infect Dis. 1991 Jun;163(6):1348-51. doi: 10.1093/infdis/163.6.1348. PMID 1645385
- [Background] Jacobson MA, Gambertoglio JG, Aweeka FT, Causey DM, Portale AA. Foscarnet-induced hypocalcemia and effects of foscarnet on calcium metabolism. J Clin Endocrinol Metab. 1991 May;72(5):1130-5. doi: 10.1210/jcem-72-5-1130. PMID 1827127
- [Background] Jacobson MA, Wulfsohn M, Feinberg JE, Davis R, Power M, Owens S, Causey D, Heath-Chiozzi ME, Murphy RL, Cheung TW, et al. Phase II dose-ranging trial of foscarnet salvage therapy for cytomegalovirus retinitis in AIDS patients intolerant of or resistant to ganciclovir (ACTG protocol 093). AIDS Clinical Trials Group of the National Institute of Allergy and Infectious Diseases. AIDS. 1994 Apr;8(4):451-9. doi: 10.1097/00002030-199404000-00006. PMID 8011248
- [Background] Reddy MM, Grieco MH, McKinley GF, Causey DM, van der Horst CM, Parenti DM, Hooton TM, Davis RB, Jacobson MA. Effect of foscarnet therapy on human immunodeficiency virus p24 antigen levels in AIDS patients with cytomegalovirus retinitis. J Infect Dis. 1992 Sep;166(3):607-10. doi: 10.1093/infdis/166.3.607. PMID 1323624
- [Background] Farese RV Jr, Schambelan M, Hollander H, Stringari S, Jacobson MA. Nephrogenic diabetes insipidus associated with foscarnet treatment of cytomegalovirus retinitis. Ann Intern Med. 1990 Jun 15;112(12):955-6. doi: 10.7326/0003-4819-112-12-955. No abstract available. PMID 2160217